CLINICAL TRIAL: NCT05124262
Title: Effect of a Low- Fermentable-Oligo-Di-Monosaccharides and Polyols (FODMAPs) Diet Group Intervention on IBS Symptoms and Fatigue
Brief Title: Effect of a Low- Fermentable-Oligo-Di- Monosaccharides and Polyols Diet Group Intervention on IBS Symptoms and Fatigue
Acronym: FODMAPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Aleris Gastromottagningen City (Unknown)
Responsible Party: Principal Investigator, Perjohan Lindfors, Operations Manager and Chief Physician, Karolinska Institutet
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GMC-FODMAPgroup
Record Dates: First submitted 2021-10-26; First posted 2021-11-17 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: Low FODMAPdiet
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with direct or delayed treatment start
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-FODMAPdiet group (Experimental): Low-FODMAPdiet intervention as group treatment in three steps during 12 weeks, elimination, re-introduction and personalization of the diet. This group of participants starts immediate.
  Interventions: Other: Low- FODMAPdiet group intervention
- Delayed start of treatment low-FODMAPdiet group (Experimental): Delayed start of treatment. This arm starts after three months
  Interventions: Other: Low- FODMAPdiet group intervention

INTERVENTIONS:
Other: Low- FODMAPdiet group intervention — Diet intervention

SUMMARY:
Irritable bowel disease (IBS) is a functional gastrointestinal disorder that affects 10% of the population. Comorbidities are common and fatigue is the most common extraintestinal complaint in IBS patients. There are no cure for the disease but there are nutrition treatments that can relieve symptoms. The main goal of this randomized controlled trial is to test the hypothesis that low-Fermentable- oligo-di- monosaccharides and polyols (FODMAPs) diet kan decrease gastrointestinal symptoms and improve quality of life and fatigue in patients with IBS.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a functional gastrointestinal disorder characterized by stomach pain at least one day a week accompanied by change in stool frequency or appearance. Prevalence of IBS is about 10 % of the population worldwide and more common in women. IBS is divided into different subclasses: diarrhea predominant, (IBS-D), predominant constipation, (IBS-C), mixed bowel habits, (IBS-M). Comorbidities are common and fatigue is the most common extraintestinal complaint among the patients. Patients has severely reduced quality of life, reduced work capacity and the cost are substantial for the patients and the society. IBS can´t be cured but the symptoms can be relieved by pharmacological as well as non-pharmacological treatment as psychological- and nutritional treatment. The main goal of this randomized controlled trial is to test the hypothesis that low FODMAPdiet kan decrease gastrointestinal symptoms and improve quality of life and fatigue in patients with IBS.

FODMAPs is an acronym for Fermentable-Oligo-Di-Monosaccharides and Polyols. FODMAPs are carbohydrates that can't be absorbed/splinted in the large intestine and they ferment rapidly and exacerbate gastrointestinal symptoms as flatulence, pain, bloating and loose stools. In total 120 patients with IBS-D and IBS-M will be randomized to immediate treatment start or delayed treatment start. The treatment will be performed in clinical setting, led by a dietitian and in group format including 12 patients in each group. The intervention time is 12 weeks with 5 group visits at a gastroenterology unit. The low-FODMAP treatment is divided into three steps: elimination of FODMAPs, re-introduction and personalization of the diet. Compliance to the diet will be measured by monitoring the FODMAP intake from three day food diaries and a compliance form. Questionnaires will be self reported in a web based application. Food diaries and the stomach diary will be filled out at baseline, at week 5, 12 and 6, 12 and 24 months post intervention.

ELIGIBILITY:
Inclusion criteria:

* Established IBS-D by RomeIV- criteria
* Established IBS-M by RomeIV- criteria
* Body Mass Index (BMI)18-35

Exclusion criteria:

* Pregnancy
* Lactation
* Ongoing eating disorder/ contact with eating disorder unit
* Postoperative gastrointestinal surgery that may impact on the gastrointestinal function
* Celiac disease
* Psychiatric disorder
* Other disorder that may impact the possibility to participate in group treatment
* Diabetes
* Ongoing low- FODMAPdiet treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in IBS Symptom Severity Scores (IBS-SSS) | Change in baseline week 0 and after elimination at week 5, after intervention at week 12, at week 38 and at 1 year and 3 months and 2 years and three months. Within each patient.
  Visual Analogues Scale (VAS-scale), composite score measuring bloating, bowel habits, satisfaction with with bowel habits and how IBS impact on QOL. Minimum score 0 and maximum score 500, higher scores indicates more severe disease

SECONDARY OUTCOMES:
Change in Multidimensional Fatigue Inventory (MFI-20) | Between baseline week 0 and after elimination at week 5, after intervention at week 12, at week 38 and at 1 year and 3 months and at 2 years and three months. Within each patient.
  The Multidimensional Fatigue Inventory-20 (MFI-20) assesses 5 dimensions of fatigue, the severity of general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue. Each dimension contain 4 questions. In total 20 questions. Minimum score 0 and maximum score 100. A higher score indicate more severe fatigue.
Change in the gastrointestinal symptom rating scale (GSRS-IBS) | Between baseline week 0 and after elimination at week 5, after intervention at week 12, at week 38 and at 1 year and 3 months and at 2 years and three months. Within each patient.
  Measuring gastrointestinal symptom severity. Contains 13 questions. Minimum score 13 and maximum score 91. Higher score indicate more severe gastrointestinal symptoms.
Change in Visceral sensitivity index (VSI) | Baseline week 0 and after intervention at 12 weeks and at week 38 and at 1 year and 3 months and 2 years and three months. Within each patient.
  The VSI questionnaire measures GI-specific anxiety, and it includes the cognitive, affective, and behavioral response to fear of GI symptoms, and the context in which these occurs. The questionnaire contains 15 questions. Minimum score 0 and maximum score 75. A higher score indicates a more severe gastrointestinal anxiety.
Change in Sickness behaviour (SQ) | Baseline week 0 after intervention at 12 weeks and at week 38, at 1 year and 3 months and 2 years and three months. Within each patient.
  Measuring symptoms that occur after acute or chronic inflammation/ infection ie. malaise, listlessness, inability to concentrate, depressed mood and lack of interest in food and surroundings. The form contains 10 questions. Minimum score 0 and maximum score 30. Higher score indicates more severe sickness behaviour.
Change in World Health Organisation (WHO) Disability Assessment Schedule (WHODAS 2.0) | Baseline week 0 and at 12 weeks and at week 38, at 1 year and 3 months and 2 years and three months. Within each patient.
  Measuring difficulties due to state of health. 12 questions. Minimum score is 12 and maximum score is 48. Higher score indicates more severe difficulties due to state.

OTHER OUTCOMES:
Change in three day food diary measuring FODMAPintake for compliance to diet intervention | Baseline week 0, after intervention at 12 weeks and at 38 weeks, at 1 year and three months at 2 years and three months.. Within each patient.
  Patient report food intake during three days. Two weekdays and one saturday or sunday.
Change in meal pattern stomach diary 7 days, | Baseline week 0, after intervention at 12 weeks and at 38 weeks, at 1 year and three months and at 2 years and three months. Within each patient.
  Measuring meal pattern
Change in stool pattern stomach diary 7 days | Baseline week 0, after intervention at 12 weeks and at 38 weeks, at 1 year and three months and at 2 years and three months. Within each patient.
  Measuring stool pattern
Change in compliance to FODMAP intervention and level of introduction of FODMAPs | Postintervention at 12 weeks and at 38 weeks, 1 year and three months and at 2 years and three months. Within each patient.
  Patients selfreport if they have reintroduced the different FODMAPs ie. fructose, lactose, fructan, galactooligosaccharides and polyols.
Change in Generalized Anxiety disorder (GAD-7) | Baseline week 0 and after 1 year and three months. Within each patient.
  Measuring anxiety in total 7 questions added with questions about how the anxiety impacts your life. Minimum score 7 and maximum score 28. Higher score indicate more severe anxiety.
Change in Patients Health questionnaire (PHQ-9) | Baseline week 0 and at 1 year and three months. Within each patient.
  Screening for depressive symptoms. 9 questions. Minimum score 0 and maximum score 27.

CONTACTS AND LOCATIONS:
Overall Officials: PerJohan Lindfors, MD, Med. dr, Principal Investigator — Karolinska Institutet